CLINICAL TRIAL: NCT04559633
Title: Anxious School Refusal in Adolescents: Efficiency of a Cognitive and Behavioral Therapy (CBT) Day Hospital Program
Brief Title: Cognitive and Behavioral Therapy in School Refusal
Acronym: RSA-Coll
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL20_0048
Record Dates: First submitted 2020-08-18; First posted 2020-09-23 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-05

CONDITIONS: Child Psychiatry; Adolescent; Anxious School Refusal; Cognitive Behavioral Therapy
Keywords: Anxious school refusal; anxiety disorders; CBT; treatment outcome; adolescents
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anxious school refusal (Experimental): Adolescents with anxious shool refusal will beneficiate of cognitive and behavioral therapy (CBT) in order to help them to return back to school
  Interventions: Other: cognitive and behavioral therapy (CBT)

INTERVENTIONS:
Other: cognitive and behavioral therapy (CBT) — The CBT program is delivered by a multidisciplinary team with 4 half day hospitalization that includes individual, group CBT and education time (2 hours per day delivered by the teacher). Participants have homework to do in their own time at home.
  CBT is a manualized program with anxiety psychoeducation, stress management, cognitive restructuration, problem solving techniques, progressive exposure, assertiveness exercises and self-esteem work.

SUMMARY:
Anxious school refusal (ASR) is a common disorder which concerns more and more adolescents who are at worse completely absent from school. A specific ambulatory cognitive and behavioral therapy (CBT) program has been established to gradually reintegrate the child back into the school environment with a multidisciplinary team. Alongside school reintegration assessment, the child's overall ability to function and anxiety levels will be measured before and after the program with additional assessments made after a further 6 and 12 months have elapsed.

DETAILED DESCRIPTION:
ASR concerns children and adolescents who feel anxiety about going to school. Some are totally absent, some just have difficulty remaining in school for the entire day, or go to school following behavioral problems such as morning tantrums or psychosomatic complaints. Anxiety disorders are the main diagnostic underlying this behavioral problem, with one or many anxiety disorders associated (i.e. separation anxiety disorder, panic disorder, social anxiety disorder, generalized anxiety disorder or specific phobia). ASR causes much distress to the child, the parents, and the school personnel and interferes with social and educational development. Children with severe or chronic school refusal appear to have a long-term risk of adult mental health issues (e.g. anxiety, depression). Studies about ASR are few, and nonexistent in France. ASR occurs in approximately 1% of all school-aged children, and 5% of all clinic-referred children, is equally common in both boys and girls but more frequent in adolescents. Recommendations for anxiety disorder treatment in youth is psychotherapy. CBT, especially exposure-based, is the intervention that is supported by numerous, randomized, controlled trials in this area. But concerning ASR, there are few studies.

A specific ambulatory therapeutic CBT program for totally absent from school adolescents is established within the children and adolescent psychiatric unit in the University Hospital of Montpellier, France. The unit has implemented CBT techniques to gradually reintegrate the child back into the school environment. This program will be implemented in 3 other child and adolescent psychiatry centers (Marseille, Béziers and Nîmes).

The main objective of this study is to evaluate the efficiency of a CBT program on the return back to school.

Secondary objectives are:

1. To evaluate the feasibility in implantation of this program
2. To describe the characteristics of adolescents
3. To assess the initial severity of mental disorders and the evolution of these disorders
4. To describe the evolution of patient anxiety
5. To describe the evolution of the overall functioning
6. To evaluate the efficiency on the return back to school at 6 and 12 month after intervention.

ELIGIBILITY:
Inclusion criteria:

* Adolescents between 10 and 16 years old registered in French college (6è to 3è),
* Anxious school refusal based on Berg's criteria,
* Completely dropped out from school (>5 consecutive days of school nonattendance, absenteeism < 12 months),
* Anxiety disorder as a principal diagnosis (DSM 5)(MINI -S KID),
* Adolescents want to return to school,
* Signed consent by parents and adolescents

Exclusion criteria:

* Intellectual disabilities
* Autism spectrum disorder
* Learning disabilities that causes emotional trouble and being the primary cause of teenagers dropping out of school.
* Conduct disorder (DSM 5)
* Ongoing psychotherapeutic care that the parents or the adolescent would not wish to suspend
* Participation in other ongoing research
* Pregnancy
* Patient not benefiting from a social security scheme

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
School continue reintegration | 46 months
  The return back to school next year : school continue reintegration (number of hours the adolescent attended school > 80% of the number of hours expected for each patient

SECONDARY OUTCOMES:
Types of anxiety disorders according to the DSM 5 | 46 months
  The questionnaire Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-S KID) is completed with parents and the adolescent
Presence of comorbidities | 46 months
  Presence of comorbidities is evaluated by the questionnaire Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-S KID) completed with parents and the adolescent
Initial severity of mental disorders and the evolution of these disorders | 46 months
  Mesure thanks to the Clinical Global Impression (CGI) scale.
Anxiety assessment | 46 months
  Mesure thanks to the Anxiety and Phobia Behavioural (ECAP) Scale
Anxiety assessment | 46 months
  Mesure thanks to the scales Revisited Children's Manifest Anxiety scale (RCMAS)
Anxiety assessment | 46 months
  Mesure thanks to the scales Multidimensional Anxiety Scale for Children (MASC)
Global functioning | 46 months
  Mesure thanks to the scale Children's global Assessment (C GAS) Scale
School attendance time month by month | 46 months

CONTACTS AND LOCATIONS:
Overall Officials: Hélène DENIS, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No